CLINICAL TRIAL: NCT04658095
Title: A Prospective, Randomized, Multicenter Study To Compare The Safety And Effectiveness Of The OMNI® Surgical System And The iStent Inject In Pseudophakic Eyes With Open Angle Glaucoma. The TRIDENT European Trial
Brief Title: Study of OMNI Surgical System and iStent for Eyes With OAG (Trident)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07062
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Ab-interno canaloplasty and trabeculotomy using the OMNI Surgical System (Active Comparator): Sequential canaloplasty (up to 360 degrees) and trabeculotomy (up to 360 degrees)
  Interventions: Device: Canaloplasty and trabeculotomy with the OMNI system.
- Ab-interno canaloplasty (360 degrees) using the OMNI Surgical System (Active Comparator): Canaloplasty alone (up to 360 degrees)
  Interventions: Device: Canaloplasty
- Ab-interno implantation of iStent inject (2 microstents) (Active Comparator): Implantation of trabecular micro bypass stents as per manufacturer's instructions.
  Interventions: Device: iStent inject

INTERVENTIONS:
Device: Canaloplasty and trabeculotomy with the OMNI system. — Ab-interno canaloplasty (360 degrees) and up to 360 degrees trabeculotomy
  Arms: Ab-interno canaloplasty and trabeculotomy using the OMNI Surgical System
Device: iStent inject — Ab-interno implantation of iStent inject (2 microstents)
  Arms: Ab-interno implantation of iStent inject (2 microstents)
Device: Canaloplasty — Ab-interno canaloplasty (360 degrees) using the OMNI
  Arms: Ab-interno canaloplasty (360 degrees) using the OMNI Surgical System

SUMMARY:
First, to compare safety and effectiveness outcomes for canaloplasty and trabeculotomy using the OMNI Surgical System to implantation of the iStent inject in lowering intraocular pressure (IOP) in pseudophakic eyes with open angle glaucoma (OAG), and second, to compare safety and effectiveness outcomes for canaloplasty alone (using the OMNI Surgical System)to implantation of the iStent Inject in lowering IOP in pseudophakic eyes with OAG.

DETAILED DESCRIPTION:
A multicenter, prospective, parallel group study planned to randomize 459 subjects to either 1)canaloplasty + trabeculotomy with the OMNI, 2)canaloplasty alone with the OMNI, or 3)iStent inject in an equal allocation ratio (1:1:1); The study includes baseline and terminal (Month 12) washout. Up to 26 centers in the UK and EU were planned to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 years or older
2. Pseudophakic
3. Diagnosis of open angle glaucoma (OAG)
4. On 1-5 ocular hypotensive medications

Exclusion Criteria:

1. Any of the following prior treatments for glaucoma:

   * Suprachoroidal stent (e.g. Cypass, iStent Supra)
   * Laser trabeculoplasty ≤ 8 weeks prior to Baseline visit with a MIGS or other glaucoma device including but not limited to iStent, iStent inject, Hydrus, CyPass
   * Trabeculectomy or other bleb forming procedure including Xen, PreserFlo, Express, glaucoma draining device/valve
   * Prior canaloplasty, goniotomy, or trabeculotomy including procedures with GATT, Kahook Dual Blade, iTrack, Trabectome
   * Ciliary ablation procedures including Endocyclophotocoagulation (ECP), Cyclophotocoagulation (G probe), Micropulse laser, or high intensity focused ultrasound (HIFU)
2. Any other form of glaucoma other than OAG
3. Concurrent ocular pathology or systemic medical condition which, in the Investigator's judgment, would either place the subject at increased risk of complications, contraindicate surgery, place the subject at risk of significant vision loss during the study period (e.g., wet AMD, corneal edema, Fuch's dystrophy, active intraocular infection or inflammation within 30 days prior to Screening Visit, etc.), or interfere with compliance to elements of the study protocol (e.g., returning to investigator's office for follow-up visits).
4. Women of childbearing potential if they are currently pregnant or intend to become pregnant during the study period; are breast-feeding; or are not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Dickerson, PhD, Study Director — Sight Sciences, Inc.
Locations (5):
- BurgerHospital, Frankfurt, Germany
- Spain (3):
  - Institut Catala de Retina (ICR), Barcelona
  - Universidad Complutense de Madrid, Valencia
  - Paseo Isabel la Católica 1-3. Edificio general Hospital Miguel Servet. Planta calle, Zaragoza
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Canaloplasty Only With the OMNI Surgical System: Subjects randomized to canaloplasty only with the OMNI surgical system
- Canaloplasty + Trabeculotomy With the OMNI Surgical System: Subjects randomized to canaloplasty and trabeculotomy with OMNI
- iStent Inject: Subjects randomized to iStent inject
Period: Overall Study
Arm/Group | Canaloplasty Only With the OMNI Surgical System | Canaloplasty + Trabeculotomy With the OMNI Surgical System | iStent Inject
Started | 5 | 1 | 4
Completed | 0 | 0 | 0
Not Completed | 5 | 1 | 4
Not completed — Study terminated | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis population will contain all subjects for whom either the OMNI (canaloplasty alone), OMNI (canaloplasty AND trabeculotomy), or iStent inject is attempted.
  The study was terminated early due to a business decision.
Groups:
- OMNI-Canaloplasty Only: All subjects for whom the OMNI (canaloplasty alone) is attempted
- OMNI-canaloplasty + Trabeculotomy: All subjects for whom the OMNI (canaloplasty+trabeculotomy) is attempted
- iStent Inject: All subjects for whom the iStent inject is attempted
- Total: Total of all reporting groups
Arm/Group | OMNI-Canaloplasty Only | OMNI-canaloplasty + Trabeculotomy | iStent Inject | Total
Number analyzed (Participants) | 5 | 1 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (3.5) | 71 (0) | 74.5 (5.1) | 74.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 5
  Male | 3 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 1 | 3 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 1 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 | 0 | 1 | 2
  Spain | 4 | 1 | 2 | 7
  Poland | 0 | 0 | 1 | 1
Diurnal IOP (DIOP) [Mean (Standard Deviation); unit: mm Hg] — Diurnal IOP is the mean of IOP measurements taken at 9AM, noon, and 4PM using Goldmann tonometry. The baseline DIOP is assessed after subjects have gone through a glaucoma medication washout.
  mm Hg | 29.0 (4.4) | 26 (0) | 24.3 (0.5) | 26.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Unmedicated DIOP From Baseline at the 12-month Postoperative Examination
Description: Mean change in unmedicated DIOP from baseline at the 12-month postoperative examination is the mean of the difference between the baseline DIOP and the Month 12 DIOP for each subject. Baseline and Month 12 DIOP are measured after appropriate washout of any glaucoma medications.
Time Frame: 12 months
Population: Results are not presented for this outcome as no subjects had reached the primary endpoint of Month 12 at the time of study termination.
Groups:
- Canaloplasty Only: Subjects randomized to canaloplasty only with the OMNI surgical system
- Canaloplasty + Trabeculotomy: Subjects randomized to canaloplasty + trabeculotomy with the OMNI surgical system
Arm/Group | Canaloplasty Only | Canaloplasty + Trabeculotomy | iStent Inject
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- OMNI-canaloplasty Alone: The safety analysis population will contain all subjects for whom the OMNI (canaloplasty alone) is attempted
- OMNI-canaloplasty + Trabeculotomy: The safety analysis population will contain all subjects for whom the OMNI (canaloplasty+trabeculotomy) is attempted
- iStent Inject: The safety analysis population will contain all subjects for whom the iStent injectis attempted
Arm/Group | OMNI-canaloplasty Alone | OMNI-canaloplasty + Trabeculotomy | iStent Inject
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 1/1 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMNI-canaloplasty Alone (N=5) | OMNI-canaloplasty + Trabeculotomy (N=1) | iStent Inject (N=4)
IOP elevation (Eye disorders) | 2 (2) | 0 (0) | 0 (0) — IOP elevation. Both AE occurred in subject study eye; Both subjects randomized to canaloplasty
Anterior chamber inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Anterior chamber inflammation - Occurred in study eye; subject randomized to canaloplasty.
Allergic conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Allergic conjunctivitis (non-infectious) - occurred in study eye. Subject randomized to canaloplasty.
Tendinitis (General disorders) | 1 (1) | 0 (0) | 0 (0) — Tendinitis-right tibialis,anterior, n (%). Subject randomized to canaloplasty.
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — COVID-19. One subject in canaloplasty arm, one subject in canaloplasty+trabeculotomy arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's publication of trial results, the Institution and Principal Investigator may publish the results of the Study generated by the Institution, subject to the obligations of the CTA, and prior approval of Sponsor in writing. The Institution shall furnish Sponsor with a written copy of any proposed publication or disclosure at least 60 days prior to submission for publication or disclosure. Sponsor may request changes or other measures to ensure the information is fairly stated.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04658095/Prot_SAP_000.pdf